CLINICAL TRIAL: NCT05173636
Title: Effects of Cervical Lateral Glide Mobilizations Along With Thoracic Mobilizations in Patients With Neurogenic Cervicobrachial Pain.
Brief Title: Effects of Cervical Lateral Glide Along With Thoracic Mobilizations in Patients With Neurogenic Cervicobrachial Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01051 Alisha Khan
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Cervicobrachial Syndrome
Keywords: Pain; Range of motion; Cervicobrachial pain; Cervical lateral glide; Thoracic mobilization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical lateral glide (Experimental): A cervical segmental contralateral lateral glide treatment technique is performed at 1 or more motion segments of the cervical spine (C5-T1), including the level(s) of the segmental motion restriction. With the patient in a supine position, the therapist cradled the head and neck above, and including, the level to be treated and performed a lateral translatory movement away from the involved side while minimizing gross cervical side flexion or rotation.
  Interventions: Other: cervical lateral glide; Other: thoracic mobilization technique
- thoracic mobilization (Experimental): A posteroanterior unilateral pressure will be applied over the transverse processes at T2-T5 on the ipsilateral side of pain in prone position.
  Interventions: Other: cervical lateral glide; Other: thoracic mobilization technique

INTERVENTIONS:
Other: cervical lateral glide — A cervical segmental contralateral lateral glide treatment technique is performed at 1 or more motion segments of the cervical spine (C5-T1), including the level(s) of the segmental motion restriction. With the patient in a supine position, the therapist cradled the head and neck above, and including, the level to be treated and performed a lateral translatory movement away from the involved side while minimizing gross cervical side flexion or rotation.
Other: thoracic mobilization technique — Participants in group B will be given cervical lateral glide along with thoracic mobilization technique in prone position.

SUMMARY:
In the scientific literature, cervicobrachial pain is the presence of pain in the neck that radiates or refers to the arm. It is considered as common spine disorder with upper quadrant pain due to muscles, joints or intervertebral discs. This study aims to compare the effects of direct neural tissue technique that is cervical lateral glide mobilization along with indirect neural tissue mobilization technique that is thoracic mobilization on pain, range of motion, endurance of neck flexors and functional ability in patients with cervicobrachial pain.

DETAILED DESCRIPTION:
The exact incidence of cervicobrachial pain syndrome is not known due to the paucity of population-based studies, patients suffering the symptoms of this condition frequently attend for physiotherapy.

In the scientific literature, cervicobrachial pain is the presence of pain in the neck that radiates or refers to the arm. It is considered as common spine disorder with upper quadrant pain due to muscles, joints or intervertebral discs. Upper quadrant discomfort involves neck, shoulder, arm, upper back but neural tissue sensitivity to mechanical stimuli portrays to be the essential element of cervicobrachial pain. It generally refers to neck pain that along with paresthesia is radiating to one upper extremity and leading to muscle imbalances. Elvey planned some clinical tests to recognize the problems of neurogenic disorders that are responsive to non-intrusive physical therapy treatment. The acceptability of these tests from effective treatments has not been adequately proven yet.

According to the literature cervical lateral glide is considered as first line treatment in reducing pain and improving upper limb function and is specifically very effective in patients of cervicobrachial pain syndrome. Cervical lateral glide has hypoalgesic effect on neck and arm pain. It is thought that this technique stimulates cervical afferents which can affect pain processes at spinal cord and cortical levels. A study was conducted in which passive techniques for mobilizing neural tissue and cervical spine were given as direct manual therapy treatment. Thoracic mobilization corresponds to indirect neural mobilization that is effective in reducing pain and functional limitations when incorporated with cervical spine mobilization that is referred as direct neural mobilization in patients of cervicobrachial pain. Evidence suggests that improvement in cervical stability and thoracic mobility achieved through manual therapy is significant in reducing neck pain and improving functional motion This study would help to investigate the delineation between specific and non-specific components of manual therapy. This study aims to compare the effects of direct neural tissue technique that is cervical lateral glide mobilization along with indirect neural tissue mobilization technique that is thoracic mobilization on pain, range of motion, endurance of neck flexors and functional ability in patients with cervicobrachial pain.

ELIGIBILITY:
Inclusion Criteria:

* Pain in upper quadrant associated with cervical spine eliciting unilateral neck pain.
* Paresthesia and numbness in the neck and arm for at least three continuous months
* Active movements of cervical spine (extension, lateral flexion to either side or ipsilateral rotations) and arm movements reproducing pain.
* Symptom reproduction on passive movements in the same pattern as with active movements.
* Elicitation of adverse response (in terms of range of movement and reproduction of symptoms) to neural tissue provocation testing of median, ulnar and radial nerves and subsequent symptom alteration with neural tissue differentiating maneuvers.
* Tenderness at transverse processes of cervical spine (nerve roots), nerve trunks of median, ulnar and radial nerves at different anatomical locations in the course of respective neural tissue.
* Hyperalgesic related cutaneous tissues on palpation (tender points).
* Evidence of a related pathology (example: radiological evidence of cervical disc pathology in the vicinity of involved nerve roots or evidence of stenosis at cervical neural foramen as diagnosed by a qualified musculoskeletal Radiologist)
* provoked or spontaneous paresthesia and pain with radicular distribution
* Positive results in the following tests: Spurling, Distraction, and Upper Limb tension test.
* Diagnosis will be based upon subjective presentation of patient's pain pattern which includes somatic referred pain and neurogenic radiating symptoms.

Exclusion Criteria:

* Bilateral symptoms (due to unilateral nature of lateral glide mobilization technique).
* History of spinal surgery
* Systemic diseases besides neck pain.
* Vertebral infections.
* Presented red flags.
* Used analgesics within 48 hours before initial assessment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for pain | at base line
  Numeric pain rating scale is used to capture the patient's level of pain. Patients will be asked to indicate the intensity of current, best, and worst levels of pain over the past 24 hours using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable). This scale exhibit fair to moderate test-retest reliability and show adequate responsiveness in patients with neck pain. Assessment to be done at base line
Numeric pain rating scale for pain | at 2nd week
  Numeric pain rating scale is used to capture the patient's level of pain. Patients will be asked to indicate the intensity of current, best, and worst levels of pain over the past 24 hours using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable). This scale exhibit fair to moderate test-retest reliability and show adequate responsiveness in patients with neck pain. Assessment to be done at 2nd week.
Numeric pain rating scale for pain | at 4th week
  Numeric pain rating scale is used to capture the patient's level of pain. Patients will be asked to indicate the intensity of current, best, and worst levels of pain over the past 24 hours using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable). This scale exhibit fair to moderate test-retest reliability and show adequate responsiveness in patients with neck pain. Assessment to be done at 4th week.
Northwick Park neck pain questionnaire (for physical function) | at baseline
  Function will be measured by the Northwick Park Neck Pain Questionnaire that is divided into nine-five parts sections. The questionnaire is easy for patients to complete, simple to score and provides an objective measure to evaluate outcome in patients with acute or chronic neck pain. This questionnaire has been demonstrated to have short-term repeatability and long-term sensitivity to change. Assessment to be done at baseline.
Northwick Park neck pain questionnaire (for physical function) | at 2nd week
  Function will be measured by the Northwick Park Neck Pain Questionnaire that is divided into nine-five parts sections. The questionnaire is easy for patients to complete, simple to score and provides an objective measure to evaluate outcome in patients with acute or chronic neck pain. This questionnaire has been demonstrated to have short-term repeatability and long-term sensitivity to change. Assessment to be done at 2nd week.
Northwick Park neck pain questionnaire (for physical function) | at 4th week
  Function will be measured by the Northwick Park Neck Pain Questionnaire that is divided into nine-five parts sections. The questionnaire is easy for patients to complete, simple to score and provides an objective measure to evaluate outcome in patients with acute or chronic neck pain. This questionnaire has been demonstrated to have short-term repeatability and long-term sensitivity to change. Assessment to be done at 4th week
Cervical range of motion by Goniometer | at baseline
  cervical range of motion will be measured by using universal goniometer. It is a reliable tool for assessing cervical range of motion in a clinical setting and is cheap. Assessment to be done at baseline.
Cervical range of motion by Goniometer | at 2nd week
  cervical range of motion will be measured by using universal goniometer. It is a reliable tool for assessing cervical range of motion in a clinical setting and is cheap. Assessment to be done at 2nd week.
Cervical range of motion by Goniometer | at 4th week
  cervical range of motion will be measured by using universal goniometer. It is a reliable tool for assessing cervical range of motion in a clinical setting and is cheap. Assessment to be done at 4th week.
Deep neck flexor endurance test | at baseline
  Neck flexor endurance will be measured with deep neck flexor endurance test(Rectus Capitus Anterior, Rectus Capitus Lateralis, Longus Capitus, Longus Colli). It will be performed in a supine lying position by tucking patients chin in and lifting off table 1 inch. The examiner will look for substitution of the platysma or sterno-cleido mastoid muscle. The flexor endurance test showed good intertester and intratester reliability when two values were averaged and, thus, may represent a useful clinical tool for practitioners involved in treating and preventing neck pain. Assessment to be done at baseline.
Deep neck flexor endurance test | at 2nd week
  Neck flexor endurance will be measured with deep neck flexor endurance test(Rectus Capitus Anterior, Rectus Capitus Lateralis, Longus Capitus, Longus Colli). It will be performed in a supine lying position by tucking patients chin in and lifting off table 1 inch. The examiner will look for substitution of the platysma or sterno-cleido mastoid muscle. The flexor endurance test showed good intertester and intratester reliability when two values were averaged and, thus, may represent a useful clinical tool for practitioners involved in treating and preventing neck pain. Assessment to be done at 2nd week.
Deep neck flexor endurance test | at 4th week
  Neck flexor endurance will be measured with deep neck flexor endurance test(Rectus Capitus Anterior, Rectus Capitus Lateralis, Longus Capitus, Longus Colli). It will be performed in a supine lying position by tucking patients chin in and lifting off table 1 inch. The examiner will look for substitution of the platysma or sterno-cleido mastoid muscle. The flexor endurance test showed good intertester and intratester reliability when two values were averaged and, thus, may represent a useful clinical tool for practitioners involved in treating and preventing neck pain. Assessment to be done at 4th week.

CONTACTS AND LOCATIONS:
Overall Officials: maria khalid, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No